CLINICAL TRIAL: NCT05424900
Title: An Integrative Intervention for Preventing Children's Emotional Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oana David (Other)
Collaborators: The Executive Agency for Higher Education, Research, Development and Innovation Funding (Other)
Responsible Party: Sponsor-Investigator, Oana David, Professor Ph.D, Babes-Bolyai University
Organization: Babes-Bolyai University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REThink Preventive
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Emotional Problem
Keywords: online therapeutic game; emotional problems; prevention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REThink game (Experimental): REThink is a online therapeutic game developed by David and collaborators (2018), proved to be an efficient intervention for the reduction of emotional symptoms in children and adolescents.
  Interventions: Behavioral: Rethink game
- Monitoring (No Intervention): Participants in this arm will be monitored for a total of eight weeks, for comparison with the REThink game intervention (after four weeks).

INTERVENTIONS:
Behavioral: Rethink game — REThink is a online therapeutic game developed by David and collaborators (2018), proved to be an efficient intervention for the reduction of emotional symptoms in children and adolescents.
  Arms: REThink game

SUMMARY:
The general objective of the study is to test an online platform for the prevention of emotional disorders in children aged 8-12 without any clinical symptoms.

DETAILED DESCRIPTION:
The general objective of the study is to test an online platform for the prevention of emotional disorders in children aged 8-12 without any clinical symptoms. The game will be used by children and adolescents for a period of four weeks. Pre-test and post-test measurements will be taken.

ELIGIBILITY:
Inclusion Criteria:

* children aged 8 to 12 years
* parental consent provided
* al least one answer different than never true on the Childhood Trauma Questionnaire - Short Form (CTQ-SF; Bernstein & Fink, 1998; Bernstein et al., 2003), measuring dichotomically the presence of Emotional Neglect, Physical Neglect, Emotional Abuse, Physical Abuse

Exclusion Criteria:

* intellectual disability or physical limitations precluding the use of the online platform presence of a mental health disorder in the children or their enrolled parent

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 294 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Child emotion regulation | baseline; pre-intervention (one week before the intervention)
  The Emotion Regulation Index for Children and Adolescents (ERICA; Biesecker & Easterbrooks, 2001). The 13 items are measured on a five-point Likert scale, from 0 "strong disagreement" to 5"strong agreement" where higher scores represent better emotional regulation abilitie
Changes in child emotion regulation | post-test, one week after the intervention
  The Emotion Regulation Index for Children and Adolescents (ERICA; Biesecker & Easterbrooks, 2001). The 13 items are measured on a five-point Likert scale, from 0 "strong disagreement" to 5"strong agreement" where higher scores represent better emotional regulation abilities.
Children emotional regulation | baseline; pre-intervention (one week before the intervention)
  The Cognitive Emotion Regulation Questionnaire - Short (Garnefski & Kraaij, 2006) is an 18-item self-report scale that measures a total of nine different cognitive coping strategies, each addressed by two items.
Changes in children emotional regulation | post-test, one week after the intervention
  The Cognitive Emotion Regulation Questionnaire - Short (Garnefski & Kraaij, 2006) is an 18-item self-report scale that measures a total of nine different cognitive coping strategies, each addressed by two items.
child emotional simptoms | baseline; pre-intervention (one week before the intervention)
  SDQ - Strengths and Difficulties Questionnaire "Goodman R, Meltzer H, Bailey V (1998)
Changes in child emotional simptoms | post-test, one week after the intervention
  SDQ - Strengths and Difficulties Questionnaire, Goodman R, Meltzer H, Bailey V (1998)

SECONDARY OUTCOMES:
Children's irrational beliefs | baseline; pre-intervention (one week before the intervention)
  The Child and Adolescent Scale of Irrationality (CASI, Bernard & Cronan, 1999)
changes in Children's irrational beliefs | post-test, one week after the intervention
  The Child and Adolescent Scale of Irrationality (CASI, Bernard & Cronan, 1999)
child behavioral difficulties | baseline; pre-intervention (one week before the intervention)
  SDQ - Strengths and Difficulties Questionnaire, Goodman R, Meltzer H, Bailey V (1998) The strengths and difficulties questionnaire: "a pilot study on the validity of the self-report version. Eur Child Adolesc Psychiatry 7:125-130"
Mental health | baseline; pre-intervention (one week before the intervention)
  SDQ - Strengths and Difficulties Questionnaire, Goodman R, Meltzer H, Bailey V (1998) The strengths and difficulties questionnaire: "a pilot study on the validity of the self-report version. Eur Child Adolesc Psychiatry 7:125-130"
Changes child mental health | post-test, one week after the intervention
  SDQ - Strengths and Difficulties Questionnaire, Goodman R, Meltzer H, Bailey V (1998) The strengths and difficulties questionnaire: "a pilot study on the validity of the self-report version. Eur Child Adolesc Psychiatry 7:125-130"

OTHER OUTCOMES:
Child trauma | baseline; pre-intervention (one week before the intervention)
  CTQ - Childhood Trauma Questionnaire Bernstein, D. P., Stein, J. A., Newcomb, M. D., Walker, E., Pogge, D., Ahluvalia, T., ... & Zule, W. (2003). Development and validation of a brief screening version of the Childhood Trauma Questionnaire. Child abuse & neglect, 27(2), 169-190.
Child attachment | baseline; pre-intervention (one week before the intervention)
  The Security Scale (Kerns, Klepac, & Cole, 1996) is a 15-item measure of attachment security in children aged 8 to 12. The scale uses a "some kids... other kids..." format and asks respondents to select the degree to which they feel they are similar to the type of children they have previously selected, using a two-point Likert scale ("Really true for me" or "Sort of true for me".

CONTACTS AND LOCATIONS:
Locations (1):
- Babes-Bolyai University, Cluj-Napoca, Romania

IPD SHARING:
Plan to Share IPD: No